CLINICAL TRIAL: NCT01572506
Title: Assessing Mechanisms Accounting for Unexplained Anemia in the Elderly
Brief Title: Mechanisms Accounting for Unexplained Anemia in the Elderly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 999912109; 12-AG-N109
Record Dates: First submitted 2012-04-05; First posted 2012-04-06 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-09-19

CONDITIONS: Anemia
Keywords: Anemia; Elderly; Mechanisms; Red Cell Survival
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Age 70 and older with unexplained anemia
  Interventions: Drug: Biotin RBC survival
- Group 2 (Active Comparator): Age 70 and older with iron deficient anemia
  Interventions: Drug: Biotin RBC survival
- Group 3 (Active Comparator): Age 70 and older without anemia
  Interventions: Drug: Biotin RBC survival
- Group 4 (Active Comparator): Age 18 - 50 without anemia
  Interventions: Drug: Biotin RBC survival

INTERVENTIONS:
Drug: Biotin RBC survival

SUMMARY:
Background:

- Anemia occurs commonly and is associated with poor outcomes in the elderly. In about a third of anemia cases in older people (over age 65), the cause of anemia is unexplained. Anemia in older adults may be caused by the bone marrow's inability to produce red blood cells fast enough to replace older red blood cells that have died. Researchers want to look at unexplained anemia by studying the life span of red blood cells in younger adults and older adults. To do so, a vitamin called Biotin will be used as a marker on the red blood cells.

Objectives:

- To investigate possible causes of unexplained anemia in older people.

Eligibility:

* Individuals in the following groups:
* Men and women between 18 and 50 years of age who do not have anemia
* Men and women at least 70 years of age who do not have anemia.
* Men and women at least 70 years of age who have iron-deficiency anemia.
* Men and women at least 70 years of age who have anemia with no known cause.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have an overnight stay for the first study visit. They will provide a blood sample to which Biotin will be added. The blood sample with Biotin will then be returned to the participant. Twenty-four hours later, another blood sample will be collected.
* Participants will have up to 14 additional study visits. At each visit, blood samples will be collected to measure the amount of Biotin remaining in the blood.
* Participants may also provide a separate blood sample for genetic testing. These tests may provide more information about genetic causes of unexplained anemia.

DETAILED DESCRIPTION:
Anemia occurs commonly and is associated with adverse outcomes in the elderly. In approximately one third of anemia cases in patients over the age of 65 years, the cause of anemia is not readily apparent (unexplained anemia or UA). Of the various causes of anemia in young adults, overt hemolysis (either acute or chronic) is very uncommon. However, we speculate that older persons tend to develop a low grade hemolytic process which significantly reduces RBC survival, and when this is not adequately countered by increased bone marrow RBC production, anemia (UA) is the consequence. This hypothesis is supported by a few clinical observations. For example, red cells in patients with UA are generally not small and when the peripheral blood smear is examined microscopically, anisocytosis (varying cell size) is observed, as is typical in patients with hemolytic anemia. Similarly, UA is frequently associated with an elevated red cell distribution width (RDW) on electronic measurement. Furthermore, serum erythropoietin levels gradually rise with advancing age (1), and this would be consistent either with a smoldering hemolytic process or a decreased responsiveness to erythropoietin. To address the hypothesis that UA is due, at least in part, to shortened RBC survival, we propose to directly measure red blood cell survival and to correlate this with aspects of red blood cell physiology that may increase susceptibility to the hemolytic process.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Ambulatory, community dweller
* Age greater than or equal to 70 years or older or between the ages of 18 and 50 years.
* Able to understand English
* Able to complete study questionnaires as determined by the investigator
* Evidence for recent (within 1 year) clinical evaluation for blood loss directed by primary care physician or consultant in subjects referred with microcytic anemia or with referring laboratories indicative of iron deficiency. Furthermore, subjects found to have microcytic anemia will be eligible but will be referred to their primary doctor for evaluation of blood loss.
* Provide informed consent

EXCLUSION CRITERIA:

* Hemoglobin (Hb) less than 9 g/dL during screening
* History of red blood cell transfusion withinthe 3 month period prior to accrual to this study, or evidence for active bleeding as ascertained by medical history (e.g., persistent melena, hematuria or dysfunctional uterine bleeding).
* Patients for whom oral iron supplementation has been prescribed within the past two months. (Patients on a stable dose of oral iron for more than two months may be eligible).
* ALT or AST more than 3 times upper normal limitation of the time of screening
* B12 or folate deficiencies during screening period
* Estimated GFR less than 30 ml/min/1.73m(2)during screening period (by the 4-variable Modification of Diet in Renal Disease [MDRD] equation).
* Receiving hemodialysis or peritoneal dialysis for renal failure, or history of kidney transplant
* Use of exogenous erythropoietin during the past 3 months
* Any major surgery requiring general anesthesia within the past 3 months
* Treatment with chemotherapy or radiotherapy in the past 12 months
* Current diagnosis of active cancer, other than non-melanoma skin cancer and, stable prostate cancer
* History of blood disorders including thalassemia, sickle cell disease or myelodysplasia
* Current severe (NYHA Class III - IV) congestive heart failure or advanced chronic obstructive pulmonary disease
* Positive serum monoclonal protein and immunofixation
* Women who are pregnant or women planning to get pregnant during the duration of the study or those with a positive pregnancy test during screening
* Active infection requiring antibiotic treatment or HIV, Hepatitis B or C
* History of overt chronic inflammation, active Crohn s disease, rheumatoid arthritis, or diabetes(HbA1C greater than 7),
* Known hemolytic anemia
* History of prosthetic heart valve
* History of participation in biotinylation studies or handling biotinylated reagent products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-03-29; Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Measurement of red blood cell survival
  Directly measure red blood cell survival and to correlate this with aspects of red blood cell physiology that may increase susceptibilty to the hemolytic process

CONTACTS AND LOCATIONS:
Overall Officials: Josephine M Egan, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute of Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.

REFERENCES:
- [Background] Ershler WB, Sheng S, McKelvey J, Artz AS, Denduluri N, Tecson J, Taub DD, Brant LJ, Ferrucci L, Longo DL. Serum erythropoietin and aging: a longitudinal analysis. J Am Geriatr Soc. 2005 Aug;53(8):1360-5. doi: 10.1111/j.1532-5415.2005.53416.x. PMID 16078962
- [Background] Guralnik JM, Eisenstaedt RS, Ferrucci L, Klein HG, Woodman RC. Prevalence of anemia in persons 65 years and older in the United States: evidence for a high rate of unexplained anemia. Blood. 2004 Oct 15;104(8):2263-8. doi: 10.1182/blood-2004-05-1812. Epub 2004 Jul 6. PMID 15238427
- [Background] Artz AS, Fergusson D, Drinka PJ, Gerald M, Gravenstein S, Lechich A, Silverstone F, Finnigan S, Janowski MC, McCamish MA, Ershler WB. Prevalence of anemia in skilled-nursing home residents. Arch Gerontol Geriatr. 2004 Nov-Dec;39(3):201-6. doi: 10.1016/j.archger.2004.03.006. PMID 15381339